CLINICAL TRIAL: NCT01224028
Title: Double-blind, Randomized Placebo-controlled Clinical Trial for the Efficacy and Safety of a Calcineurin Inhibitor, Tacrolimus(Prograf Cap®) in Patients With Non-nephrotic Albuminuric, Normotensive IgA Nephropathy
Brief Title: A Study to Evaluate the Efficacy and Safety of Tacrolimus in Korean Nephropathy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRGNS-10-01-KOR
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: IgA Nephropathy
Keywords: Tacrolimus; Prograf; Calcinurin inhibitor; Albuminurea; Proteinurea; FK506
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus group (Experimental)
  Interventions: Drug: Tacrolimus
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tacrolimus — oral
  Other Names: Prograf; FK506
  Arms: Tacrolimus group
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
This study is to evaluate efficacy and safety of tacrolimus in the patients with non-nephrotic albuminuric, normotensive IgA nephropathy after 16 week treatment with tacrolimus (Prograf) or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IgA nephropathy confirmed by renal biopsy
* Serum creatinine measurement ≤1.5mg/ml or MDRD estimated GFR ≥ 45ml/min/1.73m2 (MDRD: Modification of Diet in Renal Disorder)
* UACR level between 0.3 and 3.0
* Blood pressure measurements < 130/80mmHg

Exclusion Criteria:

* Use of immunosuppressants for more than two weeks within last one month
* Concomitant use of ACE inhibitor, ARB, steroids or immunosuppressant, NDHP-CCB, diuretics, omega-3 fatty acids and its analogue & additional dietary to treat igA nephropathy (ACE: Angiotensin Converting Enzyme, ARB: Angiotensin Receptor Blocker, NDHP-CCB: Non-dihydropyridine-type Calcium Channel Blocker
* Pregnant or breast-feeding patients. Patients who plan to bear children or breast-feed during the study and within 6 month after completion of study
* Hypersensitivity to the investigational drug or macrolide agents
* Use of potassium-sparing diuretics
* Persistence of liver function abnormality more than 1 month or presence of acute active hepatitis
* Other investigational drug within last 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline UACR to mean value of UACR measured on week 12 and week 16 (UACR: Urine Albumin Creatinine Ratio) | Week 0, week 12 and week 16

SECONDARY OUTCOMES:
Proportion of subjects achieving more than 30% reduction of UACR level from baseline | Week 0 and week 16
Proportion of subjects achieving more than 50% reduction of UACR level from baseline | Week 0 and week 16
Proportion of subjects achieving more than 0.2 reduction of UACR level | Week 0 and week 16
Composite event rate achieving less than 0.2 or 50% reduction of UACR level | Week 0 and week 16
Changes of UACR measured between before the study and each visit | Week 0, week 4, week 8, week 12 and week 16
Incidence of adverse events according to subject's self-assessment, vital signs, investigator's assessment and labo-tests | Through week 16

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Seoul, South Korea

REFERENCES:
- [Derived] Kim YC, Chin HJ, Koo HS, Kim S. Tacrolimus decreases albuminuria in patients with IgA nephropathy and normal blood pressure: a double-blind randomized controlled trial of efficacy of tacrolimus on IgA nephropathy. PLoS One. 2013 Aug 19;8(8):e71545. doi: 10.1371/journal.pone.0071545. eCollection 2013. PMID 23977072